CLINICAL TRIAL: NCT02415478
Title: The Effect of Endoscopic Lung Volume Reduction Via Endobronchial Valves on Breath Muscle Power by Patients With COPD
Brief Title: Bronchioscopic Lung Volume Reduction (BLVR)
Acronym: BLVR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 14-002
Record Dates: First submitted 2015-03-20; First posted 2015-04-14 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease (COPD); endoscopic lung volume reduction; Endobronchial valve; physical capacity; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: endoscopic lung volume reduction by valves — Independent of the study, subject will get a bronchoscopy with chartis measurement in general anaesthesia. chartis measurement is a Balloon angioplasty. Balloon will be well-positioned in lung and filled by air for occlusion of lobe of the lung. System recognizes collateral ventilation of lobe of the lung via calculation of airflow resistance.
  Negative result allows the endoscopic placement of selfexpandig endobronchial valves in the subject lung. Inhale airflow will be inhibit an enclosed air and liquids can exhaust.

SUMMARY:
For patients with emphysema, lung volume reduction by insertion of endobronchial valves could be an expedient approach to improve the diaphragm function and the strength of breathing muscles. Therefore in the present study investigators intend to examine, whether the lung volume reduction by valves might improve the physical capacity and the quality of life.

DETAILED DESCRIPTION:
In line with routine explorations it is necessary to clarify whether a patient is suitable for the lung volume reduction by insertion of endobronchial valves. To address this question lung function diagnostics, 6-minutes-walk-test, blood withdrawal, CT of the thorax, lung perfusion scintigraphy and transthoracic echocardiography have to be performed.

After confirmation of the suitability for the endoscopic lung volume reduction patients who fulfill all other eligibility criteria will be educated about the aim and performance of the study by an investigator.

Following examination will be performed additional due to the study: determination of the strength of breathing muscles via sniff nasal pressure (PImax, PE max, P0.1), determination of the life quality index via St.-George-questionary and determination of the depression score via the Short Form 8 (SF-8) Health Survey.

After that endobronchial valve will be implanted and a permanent post-operative examination will be performed for 24 hours.

Three, respectively nine month after the implanting follow up exploration will be performed on the study patients. Once again the determination of the strength of breathing muscles, the life quality index via St.-George-questionary and the depression score via SF-8 will be performed to clarify an improvement of the physical capacity and the quality of life

ELIGIBILITY:
Inclusion Criteria:

* bilateral lung emphysema after CT
* previous guidelines-based therapy of COPD (including vaccinations against Pneumococcal infections and seasonal influenza)
* nicotine abstention for not less than three months, documented by CO-HB (haemoglobin) < 2%
* FEV 1 (Forced Expiratory Volume 1 / one second capacity) ≤ 45% of reference value, after bronchodilatation
* total lung capacity (TLC) ≥ 100% of reference value
* residual volume (RV) ≥ 175% of reference value
* patient's suitability for endoscopic lung volume reduction according to multidisciplinary decision of pneumology and thorax surgery division.
* signed Informed Consent
* understanding of the nature, significance and implications of the study
* ability to understand and follow instructions of the study stuff

Exclusion Criteria:

* echo-cardiographic right ventricular pressure (PAPsys) > 50 mmHg
* indication for a permanent anticoagulation therapy (besides ASS)
* pulmonal cachexia
* pregnancy and lactating
* permanent treatment with > 20 mg Prednison per day
* hospitalisation due to a COPD-exacerbation in the last 3 months
* > 3 steroid-treated exacerbations in the last year
* Increase of FEV1 (Forced Expiratory Volume) ≥ 20% after bronchodilatation
* severe diffusion impairment (DLCO < 20%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with severe COPD (GOLD stage III or IV)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Breath Muscle Power | Change of breathing strength 3 (respectively 9) months after the bronchoscopy
  Maximal Inspiratory Pressure (PImax)
Breath Muscle Power | Change of breathing strength 3 (respectively 9) months after the bronchoscopy
  Maximal Expiratory Pressure (PEmax)
Breath Muscle Power | Change of breathing strength 3 (respectively 9) months after the bronchoscopy
  Neuromuscular drive (P0.1)
Breath Muscle Power | Change of breathing strength 3 (respectively 9) months after the bronchoscopy
  Sniff nasal pressure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, Univ.-Prof., Principal Investigator — RWTH University Hospital MK1
Locations (1):
- RWTH Univerity Hospital, Department of Cardiology, Pneumology, Vascular Medicine and Intensive Care Medicine, Aachen, Germany